CLINICAL TRIAL: NCT06118970
Title: Impaired Decision-making Capacity in Patients Suffering From Fibromyalgia: a Cross-sectional Study
Brief Title: Reduced Ability to Make Decisions: a Study That Observe Differences in Patients With Fibromyalgia and Healthy Control
Status: Recruiting | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Andrea Polli, postdoctoral researcher, Vrije Universiteit Brussel
Other Study IDs: DeMa_FM_P01
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Decision making; Stroop task; Iowa gambling task
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with fibromyalgia syndrome: Patients with fibromyalgia will be recruited at the UZ hospital in Brussels, at local patient organisations (e.g. VLFP), at the Vrije Universiteit Brussel and via social media alerts.
  This syndrome must be confirmed by a medical diagnosis. Participants should be able to understand English, Dutch or French, they must have signed an in-formed consent and they must be at least 18 years old. Patients with other diagnoses will be excluded from this study (e.g., osteoarthritis, rheumatoid arthritis, post-cancer pain, as well as patients with primary psychiatric/neurological conditions or psychopathological disorders). Subjects with a history of substance abuse or pathological gambling and individuals with color blindness will also be excluded.
  Interventions: Other: Neuropsychological tasks and self-report questionnaires
- Healthy controls: Healthy controls will be recruited through the University of Brussels or through social media alerts. Their exclusion criteria included, in addition to those specified for the fibromyalgia group, those who were suffering from fibromyalgia or had a severe rheumatic illness. Subjects should not have pain currently or have a recent history of pain (within the past 3 months).
  Interventions: Other: Neuropsychological tasks and self-report questionnaires

INTERVENTIONS:
Other: Neuropsychological tasks and self-report questionnaires — Being a cross-sectional observational study, no intervention will be administered. Subjects will be assessed with neuropsychological tasks and self-report questionnaires.

SUMMARY:
The literature has identified impairments in various cognitive functions, including learning, memory, attention, psychomotor speed, executive function, and working memory. However, only a few studies to date have investigated impairment in the decision-making process.

The aim of this study is to evaluate decision-making skills in a group of patients with fibromyalgia and compare these results with a group of healthy controls. Specifically, investigators will evaluate four hypotheses:

1. Patients with fibromyalgia may show disadvantageous decision-making in contexts of emotional decision-making and may persevere more in their wrong choices. For this reason, investigators hypothesize that patients with fibromyalgia will more frequently choose the disadvantageous decks than the healthy control group in the Iowa Gambling Task.
2. Secondly, investigators hypothesize that patients with fibromyalgia need more time to make their choice. Consistent with this hypothesis, researchers expect to find significant differences in the average time taken by the participant to make a choice in the Iowa Gambling Task.
3. The third hypothesis is that patients with fibromyalgia may have greater difficulty inhibiting automatic responses, which may lead to longer reaction times in the Stroop task. Investigators also hypothesize that stimuli with negative emotional valence (related to the typical pain experience in fibromyalgia) may have a greater effect on patients with fibromyalgia than on healthy controls (longer reaction time in the emotional Stroop Task compared to healthy controls).
4. Finally, investigators hypothesize that anxiety, depression, sleep quality, pain, decision-making style and social support may be related to worse performance in ability-based tasks.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia syndrome (confirmed by a medical diagnosis);
* Able to understand English, Dutch or French;
* Signed an informed consent.

Exclusion Criteria:

* Other diagnoses (osteoarthritis, rheumatoid arthritis, post-cancer pain, as well as patients with primary psychiatric/neurological conditions or psychopathological disorders);
* History of substance abuse or pathological gambling;
* Color blindness;
* Not have pain currently or have a recent history of pain (ONLY FOR HEALTY CONTROL GROUP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents in Belgium and Brussels, individuals belonging to fibromyalgia patient associations (e.g. VLFP), patients being treated at the UZ hospital in brussels in brussels.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Iowa gambling task (IGT) | Baseline (cross sectional)
  This task is designed to assess cognitive function in emotional decision-making. It is a computerized decision-making task that involves uncertainty, risk assessment, and the evaluation of both reinforcement and punishment.

SECONDARY OUTCOMES:
Stroop task and Emotional Stroop task | Baseline (cross sectional)
  The Stroop test is an instrument for assessing executive functions and aims to measure an individual's ability for selective attention, cognitive flexibility, and inhibition of automatic answers.
  The Stroop task can also be manipulated to examine how emotional stimuli disrupt colour-naming performance (Emotional Stroop task).

OTHER OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | Baseline (cross sectional)
  The FIQ is a solid, worldwide-used questionnaire with a history of 20 years consisting of three domains (functional domain, physical symptom domain, and mental symptom domain). It is composed of 10 questions. The first question contains 11 items related to the ability to perform large muscle tasks - each question is rated on a 4 point Likert type scale. Items 2 and 3 ask the patient to mark the number of days they felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. Items 4 through 10 are horizontal line-ar scales marked in 10 increments on which the patient rates work difficulty, pain, fatigue, morn-ing tiredness, stiffness, anxiety and depression.
  The internal consistency of the FIQ is high (Cronbach's Alpha> 0.80). The scale is translated and validated in French and Dutch.
The Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline (cross sectional)
  The MSPSS assess an individual's perception of the social support he or she receives from family, friends, and significant others. It is a self-report measure and contains 12-items, rated on a 7-point Likert-type scale, ranging from 1 "very strongly disagree" to 7 "very strongly agree." The scale was divided into 3 subscales: family, friends, and significant other, with each section consisting of 4 items. The scale reports the three subscale scores and an overall total score. The average item rating is reported as the score for the subscales and for the total score.
  The internal consistency of the MSPSS is excellent (Cronbach's Alpha > 0.89). The scale is translated and validated in French and Dutch.
Brief Pain Inventory (BPI) | Baseline (cross sectional)
  The BPI was developed to provide a quick and easy means of measuring pain intensity and the extent to which pain interferes in the lives of the pain sufferers. Using this measure, respondents rate their worst, least, average, and current pain intensity and rate the degree to which pain inter-feres with 7 domains of functioning (general activity, mood, walking ability, normal work, rela-tions with other persons, sleep, and enjoyment of life) on a scale of 0 to 10.
  In patients with chronic non-malignant pain the internal consistency (Cronbach's Alpha) was .85 for the intensity scale and .88 for the interference scale.
  The scale is translated and validated in French and translated in Dutch.
General Decision-Making Style (GDMS) | Baseline (cross sectional)
  The GDMS was designed to assess how individuals approach decision situations. It distinguishes between 5 decision styles: a rational style, an avoidant style, a dependent style, an intuitive style and a spontaneous style. The scale consists of 25 items, each item has a score ranging from 1 to 5 (1= strongly disagree to 5= strongly agree).
  The internal consistency reliability (Cronbach's alpha) range between 0.62 and 0.84 for the five styles.
  The scale is translated and validated in French and Dutch.
Hospital Anxiety and Depression Scale (HADS) | Baseline (cross sectional)
  The HADS is a two-dimension scale developed to identify depression and anxiety among physi-cally ill patients. The HADS consists of 14 items, divided into two 7 subscales: anxiety (items reflect a state of generalized anxiety) and depression (focus on the concept of anhedonia). The respondent rates each item on a 4-point scale, higher scores indicate greater levels of anxiety or depression.
  The internal consistency of the HADS range from adequate to excellent (Cronbach's Alpha 0.67-0.93).
  The scale is translated and validated in French and Dutch.
Medical Outcomes Study Short Form 36 (SF-36) | Baseline (cross sectional)
  The SF-36 is a generic patient-reported outcome measure that quantifies health status and measures health-related quality of life. It consists of 36-item measure divided into 8 subscales and 2 composite domains. The 8 subscales are: physical functioning, role limitations due to physical problems, general health perceptions, vitality, social functioning, role limitations due to emotion-al problems, general mental health and health transition.
  The internal consistency of the SF-36 in chronic pain population is good (Cronbach's Alpha 0.76).
  The scale is translated and validated in French and Dutch.
Insomnia Severity Index (ISI) | Baseline (cross sectional)
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insom-nia. the dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime func-tioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).The internal consistency of the ISI range between good and excellent (Cronbach's Alpha 0.76 - 0.91).
  The scale is translated and validated in French and Dutch.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Polli, Researcher, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vecchio E, Lombardi R, Paolini M, Libro G, Delussi M, Ricci K, Quitadamo SG, Gentile E, Girolamo F, Iannone F, Lauria G, de Tommaso M. Peripheral and central nervous system correlates in fibromyalgia. Eur J Pain. 2020 Sep;24(8):1537-1547. doi: 10.1002/ejp.1607. Epub 2020 Jun 16. PMID 32478943
- [Background] Wu YL, Huang CJ, Fang SC, Ko LH, Tsai PS. Cognitive Impairment in Fibromyalgia: A Meta-Analysis of Case-Control Studies. Psychosom Med. 2018 Jun;80(5):432-438. doi: 10.1097/PSY.0000000000000575. PMID 29528888
- [Background] Alfeo F, Decarolis D, Clemente L, Delussi M, de Tommaso M, Curci A, Lanciano T. Decision Making and Fibromyalgia: A Systematic Review. Brain Sci. 2022 Oct 27;12(11):1452. doi: 10.3390/brainsci12111452. PMID 36358377
- [Background] Walteros C, Sanchez-Navarro JP, Munoz MA, Martinez-Selva JM, Chialvo D, Montoya P. Altered associative learning and emotional decision making in fibromyalgia. J Psychosom Res. 2011 Mar;70(3):294-301. doi: 10.1016/j.jpsychores.2010.07.013. PMID 21334501
- [Background] Cuevas-Toro AM, Lopez-Torrecillas F, Diaz-Batanero MC, Perez-Marfil MN. Neuropsychological function, anxiety, depression and pain impact in fibromyalgia patients. Span J Psychol. 2014 Nov 14;17:E78. doi: 10.1017/sjp.2014.78. PMID 26054236
- [Background] Verdejo-Garcia A, Lopez-Torrecillas F, Calandre EP, Delgado-Rodriguez A, Bechara A. Executive function and decision-making in women with fibromyalgia. Arch Clin Neuropsychol. 2009 Feb;24(1):113-22. doi: 10.1093/arclin/acp014. Epub 2009 Mar 11. PMID 19395361
- [Background] Duschek S, Werner NS, Limbert N, Winkelmann A, Montoya P. Attentional bias toward negative information in patients with fibromyalgia syndrome. Pain Med. 2014 Apr;15(4):603-12. doi: 10.1111/pme.12360. Epub 2014 Jan 21. PMID 24447855
- [Background] Fischer-Jbali LR, Montoro CI, Montoya P, Halder W, Duschek S. Central nervous activity during an emotional Stroop task in fibromyalgia syndrome. Int J Psychophysiol. 2022 Jul;177:133-144. doi: 10.1016/j.ijpsycho.2022.05.009. Epub 2022 May 16. PMID 35588963
- [Background] Mercado F, Gonzalez JL, Barjola P, Fernandez-Sanchez M, Lopez-Lopez A, Alonso M, Gomez-Esquer F. Brain correlates of cognitive inhibition in fibromyalgia: emotional intrusion of symptom-related words. Int J Psychophysiol. 2013 May;88(2):182-92. doi: 10.1016/j.ijpsycho.2013.03.017. Epub 2013 Apr 2. PMID 23557844